CLINICAL TRIAL: NCT05057065
Title: Disease Progression and Intervention of Chronic HepatitisB Based on Diabetes and Hyperlipidemia
Brief Title: A Clinical Research on Disease Progression and Intervention of Chronic HepatitisB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hong Ren (Other)
Responsible Party: Sponsor-Investigator, Hong Ren, Principal Investigator, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: LS2021037
Record Dates: First submitted 2021-09-08; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Hepatitis B, Chronic
Keywords: HBV; metabolic diseases
MeSH Terms: conditions — Hepatitis B, Chronic; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hyperlipidemia: * HBsAg(+) patients
  * TC>5.17mmol/L（200mg/dl）and（or）TG>2.3mmol/L（200mg/dl）
- diabetes: * HBsAg(+) patients
  * FPG>126 mg/dL(7.0 mmol/L)Fasting is defined as no caloric intake for at least 8 h.
- CHB without metabolic disease: * HBsAg(+) patients
  * without diabetes/ obesity/hyperlipidemia

SUMMARY:
HBV(hepatitis B virus) with metabolic comorbidities may accelerate liver disease progression and increase the risk of HCC(Hepatocellular Carcinoma)development. It is reported combination of metabolic diseases and CHB is associated with substantially increased rates of liver cirrhosis and secondary liver-related events compared to CHB alone. Consequently, hepatitis B patients with metabolic comorbidities warrant particular attention in disease surveillance and evaluation of treatment indications.

DETAILED DESCRIPTION:
Primary objective:

To evaluate the impact of metabolic disease on the progression of chronic hepatitis B

* To observe HBsAg/HBeAg/HBV DNA changes /HBsAg seroconversion
* To determine high rates of Liver Cirrhosis and Hepatocellular Carcinoma

Group 1 : CHB with diabetes Group 2 : CHB with hyperlipemia Group 3 : CHB without metabolic diseases

Study Duration (in months) 24 months

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B (positive HBsAg for at least 6 months prior to NA therapy start)
* Patients on-treatment with NAs

Exclusion Criteria:

* Treatment with immunosuppressors (including systemic corticosteroids) or anti-neoplastic treatment (including radiation therapy) <=6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.
* History of depression or uncontrolled psychiatric disorders
* Subjects protected by law or not in a position to give consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic hepatitis B patients
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of NAs therapy | 2 year
  We will follow up patients every six months and all patients with a history of hepatitis B will be tested for HBsAg(+) and HBD-DNA.The curative effect was evaluated by observing the changes of serological indexes.

SECONDARY OUTCOMES:
Incidence of liver fibrosis and cirrhosis | 2 year
  We will follow up patients every six months and all patients() with a history of hepatitis B will be tested for FibroScan. The influence of metabolic diseases on the progression of hepatitis B was evaluated by comparing the changes of liver hardness between groups（Hyperlipidemia，Diabetes and CHB without metabolic disease）

CONTACTS AND LOCATIONS:
Overall Officials: HONG REN, Prof., Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The 2nd affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No